CLINICAL TRIAL: NCT05208242
Title: Small Volume Fluid Resuscitation and Supplementation With 20% albumIn Versus Buffered Crystalloids in PatiEnts With Septic Shock
Brief Title: Strong Albumin Solutions in Patients With Septic Shock
Acronym: SWIPE2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B01459; 287590 (Other: IRAS)
Record Dates: First submitted 2021-12-13; First posted 2022-01-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Sepsis; Septic Shock; Shock, Toxic
Keywords: sepsis; septic shock; fluid therapy; hyperoncotic albumin
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: A multi-centre, randomised, open-label, feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hyperoncotic albumin (Experimental): Hyperoncotic albumin for all fluid resuscitation and also as a daily supplement, guided by daily serum albumin values, for up to 7 days.
  Interventions: Drug: hyperoncotic human albumin solution
- Buffered crystalloids (Active Comparator): Buffered crystalloid solutions for all fluid resuscitation and maintenance purposes. Participants in this arms will NOT receive any albumin during their participation.
  Interventions: Drug: Buffered crystalloid solutions

INTERVENTIONS:
Drug: hyperoncotic human albumin solution — 20% human albumin solution (presented in 100ml glass bottles)
  Arms: Hyperoncotic albumin
Drug: Buffered crystalloid solutions — Buffered crystalloids solutions for all intravenous fluid therapy
  Other Names: Hartmann's solution; Compound Sodium Lactate
  Arms: Buffered crystalloids

SUMMARY:
Sepsis is an increasingly recognised burden to healthcare systems worldwide. Intravenous fluid therapy is a common first-line intervention recommended by international guidelines. Hyperoncotic preparations of human albumin solution are widely available, but their efficacy has yet to be proven.

This randomised feasibility trial will test whether it is feasible to administer hyperoncotic albumin solutions as both fluid resuscitation and as a regular supplement in patients with early septic shock.

DETAILED DESCRIPTION:
Background to this research

Sepsis is the most severe type of infection. It happens when a patient's own immune system is trying to fight an infection, but causes damage or even failure to vital organs such as the heart, lungs or kidneys. It is a life-threatening condition and even with prompt treatment as many as 1 in 4 patients with sepsis don't survive. Septic shock is a term used to describe the worst form of sepsis, where patients need life-supporting treatments in intensive care.

Guidelines recommend doctors give fluid to patients with sepsis. This aims to improve blood flow to vital organs and reduce the risk of further damage. However, there maybe risks if patients are given too much fluid, such as developing kidney failure or even death.

Human albumin solution is a type of fluid, made from blood donated by healthy volunteers. Albumin has been used safely for many years but is more expensive compared to other fluids. Alternative fluids include solutions of salts and water that closely match the contents of human blood. Some research suggests patients with sepsis might benefit from being given albumin, particularly those with septic shock, but doctors remain unsure on whether they should give it to patients with sepsis, or whether the additional expense is worthwhile.

The overall aims of this research

The aim of this research is to test whether it is possible to give patients with early septic shock strong solutions of albumin when they arrive in intensive care. The investigators will also begin to explore the financial costs of using albumin and whether they can be justified for patients treated in the NHS.

What will happen in this research?

The investigators will conduct a study of 50 patients who are admitted to intensive care with septic shock. Patients will be randomly divided into two groups. One group will receive albumin and the other standard salt solutions. Participating patients will provide blood and urine samples shortly after their arrival in intensive care and also 2 and 5 days later. All other aspects of care and treatment will remain the same. Patients will be observed and followed up to see how they are 6 months after entering the study.

What will happen with the results?

The findings of this research will be published in a medical journal and presented at meetings where other healthcare providers can hear of our work. Every participating patient will receive a written summary of the study results. Most importantly, the results of this study will help us move forward with further research into how albumin maybe used cost-effectively in patients with sepsis in the NHS.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or documented infection
2. Organ dysfunction defined as SOFA score ≥2
3. Need for vasopressor infusion for ≥2 hours
4. Serum lactate ≥2 mmol/L
5. Eligible for critical care admission without any restrictions

Exclusion Criteria:

1. >24 hours since the time point of meeting all inclusion criteria
2. <18 years of age
3. Pregnancy
4. Patients with a known allergy to albumin
5. Jehova's witnesses or other patients expressing a known objection to the use of blood products
6. Previous receipt of human albumin solution for the episode of sepsis in question
7. Previous enrolment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
Participant recruitment rate | 24 months after opening the trial
  Evidence to confirm feasibility of the study protocol without any further modification for a future efficacy trial. This will be objectively determined by a recruitment rate of >2 participants per month, resulting in study recruitment being completed within 24 months of opening the trial. A pre-specified threshold of >80% of the anticipated recruitment rate would support the feasibility of a future efficacy trial.

SECONDARY OUTCOMES:
Vasopressor use | hourly values for up to 7-days
  The hourly use of vasopressor infusions from enrolment in mcg/kg/min
Survival | 90-days after enrolment
  Number of participants who survive
Healthcare costs | 90-days after enrolment
  Healthcare service use and costs. These will be estimated using a participant's medical records to estimate the cost of their hospital admission episode. Data on further healthcare costs will be acquired through the 90-day follow-up where participants will be asked about the healthcare service use since their discharge from hospital. All costs will be calculated in £GBP, with current equivalents in Euros and USD.
Quality of Life of study participants | 90-days after enrolment
  Healthcare related quality of life as measured by the EuroQol Research Foundation's EQ-5D-5L questionnaire via telephone. This widely validated tool assesses healthcare related quality of life across 5 domains (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each domain is scored across 5 levels, with 1 indicating 'no problems' and 5 indicating 'unable to/extreme problems'. The questionnaire also includes a self-reported health score using a visual analogue scale. This EQ-VAS derives a total health score from 0 to 100, with 100 indicating the best health a participant can imagine, and 0 indicating the worst heath imaginable.
Cumulative fluid balance (in millilitres) | daily values for up to 7 days
  This daily measure of total fluid administered minus total fluid out reflects the daily amount of fluid accumulated by participants. It will be measured on a daily basis with summary comparisons made at day 7.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Manchester Royal Infirmary, Manchester, Lancashire
  - Wythenshawe Hospital, Manchester, Lancashire

IPD SHARING:
Plan to Share IPD: No